CLINICAL TRIAL: NCT04915898
Title: Oral Care as Prevention for Non-ventilator Hospital-acquired Pneumonia: A Four-unit Cluster Randomized Study
Brief Title: Hospital-acquired Pneumonia Prevention: Intervention, Evaluation & Research
Acronym: HAPPIER-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Collaborators: Medline Industries (Industry)
Responsible Party: Principal Investigator, Daleen Penoyer, PhD,RN,CCRP,FCNS,FCCM, Director, Center for Nursing Research and Advanced Nursing Practice, Orlando Health, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18.074.06
Record Dates: First submitted 2021-02-25; First posted 2021-06-07 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Healthcare-Associated Pneumonia
Keywords: oral hygiene; non-ventilator hospital acquired pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Intervention Model Description: Cluster randomization of control and intervention groups
Who Masked: Care Provider
Masking Description: Audits on two control units with no change in oral care practices. Emphasizing that we are supporting patient hygiene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Care Hygiene Intervention Group (Active Comparator): Providing oral care kits designed to facilitate adherence to brushing teeth after meals and before sleep. Providing continuous education and feedback on performance to team members on the interventional units. Encouraging patients to brush their teeth and use the kits or own materials if desired.
  Interventions: Other: Oral Hygiene - teeth brushing
- Control group - standard of care oral care on units (No Intervention): These units will perform their 'usual' or standard of care for oral hygiene practices without use of the oral care kits, no encouragement to perform outside of usual care

INTERVENTIONS:
Other: Oral Hygiene - teeth brushing — Oral hygiene using a special kit with recommended materials and instructions: Use of an ADA approved toothbrush, toothpaste with dentifrice, antiseptic mouthwash and non-drying lip moisturizer encouraged after meals and at bedtime
  Arms: Oral Care Hygiene Intervention Group

SUMMARY:
The purpose of this study is to determine the effectiveness of a universal, standardized oral care protocol on prevention of non-ventilated hospital-acquired pneumonia (NV-HAP) in the acute care setting. In the course of the year-long study, the research team will provide educational and materials support for oral hygiene on two interventional units (one medical; one surgical) and two control units (one matched medical; one surgical). At the end of the study, the research team will evaluate existing hospital data to determine the number of NV-HAPs in the interventional and control groups.

DETAILED DESCRIPTION:
Prior to the study, the research team will have a lead-in period where education will be provided to the interventional groups and demonstration of desired oral care practices for patients (September 1-30, 2018) Design Previous research on the effectiveness of oral care for NV-HAP prevention has primarily relied on pre/post intervention study designs. In order to enhance compliance and avoid contamination of both the treatment and intervention groups, the research proposed the use of cluster randomization.

ICD-10 codes and a standardized CDC definition of non-ventilator hospital-acquired pneumonia will be used to determine the baseline incidence on NV-HAP for the 12 months prior to study implementation. The incidence will be expressed as both an overall incidence based on total patient days, as well as a rate per 1000 patient days.

The research team will follow the consolidated standards of reporting trials (CONSORT) research methods and reporting for pragmatic trials (2010). The research team will implement the HAPPI protocol using Stetler's model of implementation science. Overall the implementation process will be guided by Influencer Model ™ .

Methods There are no experimental procedures or medications use proposed in this study. The study consists of implementing a standardized oral care protocol (Attachment A) which are components of basic nursing care. Previous research has found that opportunities for oral care were often missed as part of daily care. The research team proposed to set specific standards and protocols for delivery of oral care on the intervention unit and to monitor the amount of oral care provided on both the control and intervention units.

The evidence-based oral care protocol consists of:

* oral care assessment by a RN to determine type and frequency oral care
* brushing the teeth with a soft-bristled toothbrush and plaque removing toothpaste
* rinsing with a non-alcohol based mouth wash
* application of lip and mouth moisturizer
* use of 24-hour suction toothbrush kits for high aspiration-risk patients who meet criteria, per oral care protocol

The study coordinator will provide educational information and support on the study units for use of the oral care kit and implementation of oral care after meals and before bedtime on the interventional units. As part of validation of oral care, the coordinator will make rounds on patients on the study units and validate and audit oral care activities with the patient/family and encourage their participation in oral care and with documentation checks. On the control units, the coordinator will also make rounds and evaluate oral care frequency in a non-conspicuous manner and through documentation.

ELIGIBILITY:
Inclusion Criteria:

• in-patient adults (18 and older) in control (one medical/one surgical) and interventional (one medical/one surgical) study units in whom oral care is not contraindicated

Exclusion Criteria:

* patients who are on mechanical ventilation, intubated orally, or with tracheostomy
* patients who have contraindications for oral care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8709 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Reduced non-ventilator hospital acquired pneumonia - NV-HAP | One year - October 1, 2018-September 30, 2019
  Percent reduction of hospital acquired pneumonia

SECONDARY OUTCOMES:
Incidence of NV- HAP | One year - october 1, 2018-september 30, 2019
  Incidence of NV-HAP per 1000 patient days

OTHER OUTCOMES:
Compliance to oral care practices | One year - October 1, 2018-September 30, 2019
  The number of oral care practices per patient per day

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Penoyer, PhD, RN, Principal Investigator — Orlando Health, Inc.
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No